CLINICAL TRIAL: NCT06196671
Title: Oncolytic Virus Plus PD-1 Inhibitor to Patients With Advanced Pancreatic Cancer
Acronym: PTCA199-8
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-8
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oncolytic Virotherapy; camrelizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Oncolytic virus plus PD-1 inhibitor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oncolytic virus plus PD-1 inhibitor (Experimental): * H101 intratumorally injection starts at day 1.
  * Camrelizumab will be administered at 200 mg i.v. every 3 weeks at day 2.
  * After two cycles of treatment, Camrelizumab will be administered alone at 200 mg i.v. every 3 weeks from cycle 3 until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  * The following treatment will be applied according to the newest edition of National Comprehensive Cancer Network (NCCN) guideline.
  Interventions: Drug: H101; Drug: Camrelizumab

INTERVENTIONS:
Drug: H101 — H101 15x10^11vp intratumorally injection starts at day 1.
  Other Names: Oncolytic virus
Drug: Camrelizumab — Camrelizumab will be administered at 200 mg i.v. every 3 weeks at day 2.
  Other Names: pd-1 inhibitor

SUMMARY:
The purpose of this study is to evaluate the efficacy of oncolytic virus plus PD-1 inhibitor to Patients with Advanced Pancreatic Cancer.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. In 2011, the PRODIGE trial has shown that oxaliplatin, irinotecan, fluorouracil, and leucovorin (FOLFIRINOX) was associated with a survival advantage but had increased toxicity.

Recent studies have suggested that local destruction of tumor tissue by oncolytic virus induced activation and maturation of dendritic cells and tumor-specific T cells by cross-presentation of tumor antigens. PD-1 blocking antibody interferes with PD-1 mediated T-cell regulatory signaling. Combination of PD-1 blocking antibody plus oncolytic virus may increase anti-tumor efficacy in pancreatic cancer.

The purpose of this study is to evaluate the efficacy of oncolytic virus plus PD-1 inhibitor to patients with advanced pancreatic cancer who are refractory to standard chemotherapy. Progression-free survival (PFS), objective response rate (ORR), overall survival (OS) and disease control rate (DCR) are measured every three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years and ≤ 80 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically or cytologically confirmed advanced pancreas adenocarcinoma.
* Patients who have received at least two lines of anti-tumor chemotherapy, or patients who have been unsuitable or unwilling to standard therapy.
* Locally advanced, or metastatic pancreatic cancer.
* Presence of at least of one measurable lesion in agreement to RECIST criteria.
* The expected survival ≥ 3 months.
* Adequate organ performance based on laboratory blood tests.
* Patients who are willing or able to comply with study procedures.

Exclusion Criteria:

* Pregnant or nursing women.
* Primary pancreatic cancer, or prior treatment with oncolytic virus and PD-1 inhibitor.
* The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.
* Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
* Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results.
* Allergic to study drugs.
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival，OS | At the end of Cycle 1 (each cycle is 21 days)
  OS of subjects from recruiting to the time of death from any cause

SECONDARY OUTCOMES:
progression-free survival, PFS | At the end of Cycle 1 (each cycle is 21 days)
  PFS of subjects from recruiting to the time of disease progression
objective response rate (ORR) | At the end of Cycle 1 (each cycle is 21 days)
  CR + PR
disease control rate (DCR) | At the end of Cycle 1 (each cycle is 21 days)
  CR + PR + SD

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chiu M, Armstrong EJL, Jennings V, Foo S, Crespo-Rodriguez E, Bozhanova G, Patin EC, McLaughlin M, Mansfield D, Baker G, Grove L, Pedersen M, Kyula J, Roulstone V, Wilkins A, McDonald F, Harrington K, Melcher A. Combination therapy with oncolytic viruses and immune checkpoint inhibitors. Expert Opin Biol Ther. 2020 Jun;20(6):635-652. doi: 10.1080/14712598.2020.1729351. Epub 2020 Feb 23. PMID 32067509
- [Background] Zhang Y, Qian L, Chen K, Gu S, Wang J, Meng Z, Li Y, Wang P. Intraperitoneal oncolytic virotherapy for patients with malignant ascites: Characterization of clinical efficacy and antitumor immune response. Mol Ther Oncolytics. 2022 Mar 15;25:31-42. doi: 10.1016/j.omto.2022.03.003. eCollection 2022 Jun 16. PMID 35399603